CLINICAL TRIAL: NCT02410005
Title: Kidney Disease in Type 2 Diabetes Mellitus: Biomarker Discovery and Novel Therapeutics
Brief Title: Intervention Using Vitamin D for Elevated Urinary Albumin Treated With Losartan in Diabetes (IDEAL)
Acronym: IDEAL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Logistic challenges
Sponsor: Weill Cornell Medical College in Qatar (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-00039; NPRP No: 4-1392-3-345 (Other Grant/Funding Number: Qatar National Research Fund); 14-00039 (Other: HMC/WCMC-Q JIRB)
Record Dates: First submitted 2015-02-18; First posted 2015-04-07 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Calcitriol; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan alone (Active Comparator): In the losartan alone group, subjects are prescribed: losartan 50mg twice daily.
  Interventions: Drug: Losartan
- Losartan and Calcitriol (Experimental): In the losartan plus calcitriol group, subjects are prescribed: losartan 50mg twice daily and calcitriol 0.25mcg daily.
  Interventions: Dietary Supplement: Calcitriol; Drug: Losartan

INTERVENTIONS:
Dietary Supplement: Calcitriol
  Other Names: 1,25-dihydroxycholecalciferol; 1,25-dihydroxyvitamin D3
  Arms: Losartan and Calcitriol
Drug: Losartan

SUMMARY:
This study is a single center open-label randomized controlled trial designed to evaluate the efficacy of calcitriol plus losartan therapy in subjects with type II diabetes and macroalbuminuria.

DETAILED DESCRIPTION:
The investigators propose to test the efficacy and safety of a combined regimen of calcitriol and losartan in subjects with type II diabetes (T2DM) with macroalbuminuria. Should the investigators study confirm the hypothesis that the proposed novel regimen is superior to the current practice of renin-angiotensin-aldosterone system blockade, the study would significantly advance the care of subjects with type II diabetes and kidney disease in Qatar and worldwide. In this regard it is worth noting that the prevalence of end stage renal disease in Qatar is 202 subjects per million population. This would translate into fewer subjects requiring dialysis or transplantation, an enormous benefit to individuals and society.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of T2DM requiring treatment with at least one oral hypoglycemic medication or insulin
2. Macroalbuminuria as defined as the presence of a UACR greater than 300 mg/gm creatinine (30 mg/mmol creatinine) on two occasions in the last six months
3. Estimated eGFR of 30 to 90 mL/min/1.73 m2

Exclusion Criteria:

1. Positive Pregnancy Test or planning pregnancy in the subsequent 18months (if female)
2. Serum Calcium > 2.45 mmol/L (9.8 mg/dL)
3. Serum Phosphorus > 1.78 mmol/L (5.5 mg/dL)
4. Serum Potassium > 5.5 mmol/L (5 mEq/L)
5. Parathyroid hormone < 20 pg/mL or > 500 pg/mL
6. Hemoglobin A1C > 12%
7. 25-OH Vit D > 50 ng/mL
8. Poorly controlled hypertension defined as systolic blood pressure >= 180 mm Hg or diastolic blood pressure >= 110 mm Hg
9. History of kidney stones
10. History of severe disease like chronic liver disease
11. Active malignancy
12. Active granulomatous diseases like turburculosis and sarcoidosis
13. Recent diagnosis of acute renal failure within 3 months of screening visit
14. Likelihood of renal replacement therapy within 1 year
15. History of parathyroidectomy
16. Currently taking calcitriol or 1,25-dihydroxyvitamin D analog
17. Currently taking calcitonin, bisphosphonates, cinacalcet, teriparatide, glucocorticoids or other drugs that may affect calcium or bone metabolism (subjects may be taking calcium containing phosphate binder or other phosphate binder. Subjects may also be taking stable dose of estrogen/progestin)
18. History of osteoporosis or other bone disorder requiring calcitriol therapy
19. History of allergic reaction to calcitriol, paracalcitol, hectoral, or other 1,25-dihydroxyvitamin D analogs
20. History of allergic reaction to losartan or any other angiotensin receptor blocker therapy
21. Evidence of drug or alcohol abuse

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09-07 (Actual); Study Completion 2015-09-07 (Actual)

PRIMARY OUTCOMES:
24h urine 24hr urine albuminuria | 12 month
  24h urine albuminuria (log transformed) from baseline to 12 months post-randomization in the losartan plus calcitriol group compared to the losartan alone group.

OTHER OUTCOMES:
Urine mRNA/miRNA expression | 15 months
Urine Albumin-to-Creatinine Ratio (UACR) | 15 months
Blood Pressure (BP) | 15 months
Estimated glomuerula filtration rate (eGFR) | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis August, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- Weill Cornell Medical College, New York, New York, United States
- Qatar (2):
  - Weill Cornell Medical College in Qatar, Doha
  - Hamad Medical Corporation, Doha